CLINICAL TRIAL: NCT00228670
Title: Herpesvirus in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arlene Stecenko, Principal Investigator, Emory University
Other Study IDs: IRB00041094; IPF (Other: Other)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Lung Diseases; Herpesvirus Infections
Keywords: Idiopathic Pulmonary Fibrosis; herpesvirus; lung biopsy; Having diagnosed lung disease; Scheduled to have a lung biopsy as part of the evaluation for your lung disease
MeSH Terms: conditions — Lung Diseases; Herpesviridae Infections; Idiopathic Pulmonary Fibrosis; Herpes Simplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung tissue at the time of lung transplantation. Saliva, induced sputum, and blood at clinic visitis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IPF-Clinic: Adult patients with idiopathic pulmonary fibrosis being followed in pulmonary clinic
- Controls - Clinic: Adult subjects with no underlying pulmonary disease who are the household partner of an IPF patient being followed in pulmonary clinic
- IPF-Transplant: IPF patient undergoing lung transplant
- Controls-Transplant: Lung tissue from organ donor

SUMMARY:
The purpose of this study is to: 1) to develop a method to quantify Epstein Barr Virus (EBV) load in lung tissue of humans and to determine whether EBV viral load is significantly higher in lung tissue from patients with idiopathic pulmonary fibrosis (IPF) than in control lung tissue; 2) to determine whether EBV localized to epithelial cells in IPF lungs and to relate epithelial positivity to tissue viral load; 3) to measure viral load in induced sputum from IPF subjects over time in order to determine whether periodic active herpes virus replication occurred in the respiratory tract; and 4) to compare longitudinal measures of viral load in induced sputum with simultaneously collected saliva in order to assess the clinical utility of the two approaches.

DETAILED DESCRIPTION:
IPF is a progressive disease where there is no proven treatment, other than lung transplant. Doctors do not know what causes IPF. We think that IPF is caused by a viral infection, particularly herpes virus. The goal of this experiment is to build the case for a causal link between IPF and herpes virus. This information is important to help us develop new therapies to treat patients with IPF.

We will collect lung tissue at the time of lung transplant surgery from IPF patients and from organ donors as controls. Control lung tissue was collected if it was removed as a part of regular care or would otherwise be discarded. No extra tissue was taken solely for this research project.

We will also perform a prospective longitudinal study on IPF patients and their household partners. IPF subjects are included if they have no other pulmonary disease and the diagnosis of IPF is confirmed by lung biopsy or by clinical and chest CT findings. The control group will consist of subjects without respiratory symptoms or pulmonary diseases who are the household partner or spouse of an enrolled IPF subject and who accompanies the IPF patient to outpatient clinic visits. If there is no household partner, or if the partner is unwilling to participate, we will still enroll the IPF subject who qualifies for the study and is willing to participate. Saliva, induced sputum, and venous blood will be collected from IPF and control subjects after informed consent at each clinic visit. Visits usually are at approximately 3-4 month intervals over a one year period.

ELIGIBILITY:
For the study on lung tissue, eligible subjects were IPF patients undergoing lung transplant surgery and from organ donors who died from non-pulmonary causes. For the study in clinic, subjects were IPF patients who had no other pulmonary disease other than IPF and the diagnosis of IPF was confirmed by lung biopsy or by clinical and chest CT findings. The control group consisted of subjects without respiratory symptoms or pulmonary diseases who were the household partner or spouse of an enrolled IPF subject and accompanied the IPF patient to outpatient clinic visits.

Exclusion Criteria:

* Failure of the patient to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic pulmonary fibrosis (IPF) or controls with no underlying pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2005-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Viral load | 1 year
  EBV viral load in induced sputum collected at each clinic visit over a one year period

SECONDARY OUTCOMES:
Viral load | 1 year
  EBV viral load in saliva collected every clinic visit over a one year period

OTHER OUTCOMES:
Viral load | one time point
  EBV viral load in lung tissue collected at the tim e of lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Stecenko, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States